CLINICAL TRIAL: NCT05507957
Title: Impact of Blood Culture Positivity Time on Clinical Management of Pediatric ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Salah EL-Dein Hosney, master of clincical patholofy, Assiut University
Other Study IDs: fatma elnaggar
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: direct reporting of time to positivity of blood culture to ICU to know its effect to patients managment — -Disinfection using povidone-iodine, alcohol preparation or chlorhexidine gluconate ethanol (CHG-ALC ), so that each type was used on 40 patients
  Other Names: use different type of disinfectants (povidone iodine (PVI), alcohol preparations, and chlorhexidine gluconate ethanol (CHG-ALC)

SUMMARY:
Sepsis accounts for high morbidity and mortality rates in ICU globally. Early recognition of sepsis with appropriate antimicrobial therapy is critical for the appropriate management of patients (1).

Blood culture (BC) is considered the gold standard for sepsis etiological diagnosis , with good sensitivity ,but suffering usually of delay or even failure to detect microorganisms in patients already treated with antimicrobials and failure to identify pathogens other than bacteria or yeast (2, 3).

Time-to-positivity (TTP) of blood cultures is defined as the time from the start of incubation to a positive signal. Knowledge of the distribution of blood culture TTP is of clinical benefit in the re-evaluation of patients with a clinical syndrome consistent with infection. A low probability of bacteremia when blood cultures have remained negative after 24 hours (4). Positive episodes with TTP more than or equal 24 h are commonly optimally treated infections, catheter-related infections, or infections caused by slowly growing microorganisms such as Candida or anaerobic Gram-negative bacteria. Growth of multidrug-resistant Gram-negative bacilli is exceptional beyond 24 h. In current clinical practice, bacteremia is considered unlikely if blood cultures have been negative for 48-72 hours (5, 6). Most blood culture bottles turn positive in less than 4 days, shortening the duration of incubation appears the most relevant solution in order to free additional capacity(4).

Various disinfectants, such as povidone iodine (PVI), alcohol preparations, and chlorhexidine gluconate ethanol (CHG-ALC), are used for disinfection prior to blood culture sampling. Contamination rates of cultured blood samples vary according to the disinfectant used, sampling site, definition of contamination, and skill level of individuals performing the venipuncture.(7, 8)

In this study, Investigators assessed the real life clinical impact on septic ICU patients based on time of blood culture positivity time.

DETAILED DESCRIPTION:
Aim(s) of the Research :

1. Evaluate the impact of blood culture positivity time in real -life clinical practice (patient management and reduction of ICU stay, as well as decreases in 30-days mortality.)
2. Investigates the probability of blood culture positivity after 24 hours.
3. evaluate if there was diagnostic value of TTP
4. Identify if there is difference in the blood culture contamination rate between uses of various type of disinfectant.

Sample Size Calculation: 120 septic patient in pediatric intensive care unit

Study tools:

The following will be done to all patients:

Data collection:

Clinical data (were retrieved from the medical records) :

* age and weight
* Date and time of culture collection
* pre-existing medical conditions (concomitant disease).
* Clinical parameters at presentation. The most likely source of bacteremia
* if start empirical antibiotic treatment before collection or not and its type, duration (concomitant antimicrobial therapy)
* volume of blood drawn in the bottles
* outcome data. Including change of antibiotic treatment and time to switch to directed therapy, length of ICU stay and 30-day mortality.

Microbiological data (were retrieved from the database of the Department of Medical Microbiology.) :

* date and time of bottle loading ( to know transportation time)
* date and time in which growth was first reported
* TTP(time to positivity of blood culture)
* Pathogen detected by blood culture

Blood culture sampling :

* collecting blood samples as soon as possible after the onset of clinical symptoms, ideally prior the administering antimicrobial therapy.
* Disinfection using povidone-iodine, alcohol preparation, or chlorhexidine gluconate ethanol (CHG-ALC ), so that each type was used on 40 patients
* collect 2 sets of blood culture bottles. blood culture was obtained either at one time or over a brief time period (e.g. within 1 hour) from multiple venipuncture sites.
* Blood for culture must be collected and dispensed aseptically with great care to avoid contaminating the specimen and culture medium

Blood culture handling procedures and laboratory techniques:

* Rapid transportation to microbiology unit.
* Rapid bottle loading in bioMerieux BacT/Alert Virtuo where it was incubated for 5 days
* Direct Gram stain was performed for all positive blood culture bottles.
* Followed by subculture onto solid agar media, including blood agar, chocolate agar & MacConkey agar and sabaroud agar (Diagnostic Media products(DMP). Then identification of microorganisms and antibiotic susceptibility by Vitek 2.
* Direct reporting method to the pediatric intensive care unit
* The presence of one of the following microorganisms in a single BC bottle or Blood Culture set was considered as contaminant: coagulase-negative staphylococci (CoNS), with the exception of S. lugdunensis, Propionibacterium spp., Bacillus spp. other than B. anthracis, Corynebacterium spp. (diphtheroids), Aerococcus-like organisms, Micrococcus spp., viridans group streptococci other than S. pneumoniae, and Neisseria spp. other than N. gonorrhoeae or N. meningitidis. These microorganisms were considered as significant when other BC bottles collected 48h before were positive with the same microorganism, after reviewing of clinical data.

ELIGIBILITY:
Inclusion Criteria:

* The population of our study were patients in ICU unit in pediatric hospital of Assuit University Hospitals, that presented with clinical symptoms which may lead to a suspicion of a bloodstream infection or sepsis which is:

  * Undetermined fever ( ≥ 38°C) or hypothermia ( ≤ 36°C).
  * Shock, chills, rigors
  * Severe local infections (meningitis, endocarditis, pneumonia, pyelonephritis, intra-abdominal suppuration etc.) Multiple episodes of bacteremia per patient were allowed if the antimicrobial therapy for the previous episode had been completed and clinical and microbiological cure had been achieved

Exclusion Criteria:

-blood culture bottles that were drawn in vacation days (because of no distinct control on transportation time, which affect TTP)

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The population of our study were patients in ICU unit in pediatric hospital of Assuit University Hospitals, that presented with clinical symptoms which may lead to a suspicion of a bloodstream infection or sepsis which is:
  * Undetermined fever ( ≥ 38°C) or hypothermia ( ≤ 36°C).
  * Shock, chills, rigors
  * Severe local infections (meningitis, endocarditis, pneumonia, pyelonephritis, intra-abdominal suppuration etc.)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of blood culture positivity time in patient management and reduction of ICU stay, as well as decreases in 30-days mortality. | through study completion, an average of 1 year.
  investigators measured the time to positivity of blood culture in hours. Then direct reporting the result to the physician ( as few true bloodstream infections were detected after 48 hours) ,,, Then study the impact of the result on therapeutic decisions (start of treatment, or switch or association of antibiotic/antifungal therapy). Then days of hospital stay were measured in the day unit& mortality rate was measured in percentage
Investigates the probability of blood culture positivity after 24 hours. | through study completion, an average of 1 year.
  time of positivity of blood culture measured in hours. It was calculated as the time from the start of incubation to a positive signal
evaluate if there was diagnostic value of TTP | through study completion, an average of 1 year.
  see if there was a relationship between time of positivity of blood culture (in hour unit) and the type of microorganism,, and And if TTP can distinguish between contaminant and true pathogen
Identify if there is difference in the blood culture contamination rate between uses of various type of antiseptic. | through study completion, an average of 1 year.
  Identify if there is a difference in the blood culture contamination rate (measured in percentage) between uses of various types of antiseptic.

SECONDARY OUTCOMES:
- Identify if TTP in real life was superior to expensive modern microbiological techniques for the diagnosis of sepsis | through study completion, an average of 1 year.
  expensive modern microbiological techniques for the diagnosis of sepsis are BioFire FilmArray Blood Culture Identification panel and T2 magnetic Resonance Bacterial Panel

CONTACTS AND LOCATIONS:
Overall Officials: mohammed Z Abo krisha, professor, Principal Investigator — Assiut University
Locations (1):
- Assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] endnote
- See also: Seasonal variations in blood culture numbers and time to positivity and potential impact of reducing incubation periods — https://pubmed.ncbi.nlm.nih.gov/33893569/
- See also: Time to positivity of blood cultures in patients with bloodstream infections: A useful prognostic tool — https://pubmed.ncbi.nlm.nih.gov/27916290/
- See also: Neither Blood Culture Positivity nor Time to Positivity Is Associated With Mortality Among Patients Presenting With Severe Manifestations of Sepsis: The FABLED Cohort Study — https://pubmed.ncbi.nlm.nih.gov/34307728/
- See also: Chlorhexidine alcohol versus povidone-iodine: The comparative study of skin disinfectants at the blood transfusion centers of Iran — https://pubmed.ncbi.nlm.nih.gov/32008937/